CLINICAL TRIAL: NCT06590948
Title: Clinical Application of Quantitative Major Imaging Features of Contrast-enhanced Ultrasound Liver Imaging Reporting and Data System
Brief Title: Clinical Application of Quantitative Major Imaging Features of CEUS LI-RADS
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0347
Record Dates: First submitted 2024-07-25; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Liver Cancer
Keywords: hepatic carcinoma; contrast-enhanced ultrasound; liver imaging reporting and data system; washout
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pathological results of liver masses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC
  Interventions: Diagnostic Test: contrast-enhanced ultrasound
- non-HCC
  Interventions: Diagnostic Test: contrast-enhanced ultrasound

INTERVENTIONS:
Diagnostic Test: contrast-enhanced ultrasound — contrast-enhanced ultrasound with SonoVue and quantitative analysis of liver imaging reporting and data system

SUMMARY:
Liver cancer (LC) is the sixth most common malignant tumor and the third cause of cancer mortality in the world. According to the 2018 United States Association for the Study of Liver Diseases guidelines for the diagnosis and treatment of liver cancer, patients with HCC high-risk factors can be directly diagnosed by imaging if they have typical imaging signs, without the need for puncture pathological confirmation.

Since 2011, United States the American College of Radiology (ACR) has successively launched Liver Imaging And Reporting and Data System (LI-RADS) based-on contrast-enhanced CT (CECT), contrast-enhanced MRI (CEMRI), and contrast-enhanced ultrasound (CEUS) , which have achieved good clinical diagnostic results and are constantly being updated and improved.LI-RADS provides standardized imaging diagnosis for high-risk populations and classifies each liver lesion into LR-1 to LR-5 (possibility of HCC), LR-M (probably or definitely malignant, but not HCC), LR-TIV (intravenous tumor).

Although CEUS LR-5 has a high accuracy in diagnosing HCC, there is also a considerable proportion of HCC in CEUS LR-4 and CEUS LR-3. Studies have shown that CEUS LR-M contains a high proportion of HCC, the sensitivity of CEUS LR-5 in diagnosing HCC is relatively low, and the possibility of HCC cannot be ruled out if it is not classified as CEUS LR-5. Therefore, how to improve the diagnostic sensitivity and specificity is the key goal of CEUS LI-RADS.

According to the CEUS LI-RADS diagnostic criteria, the key signs include arterial phase hyper-enhancement (APHE) and washout. The guidelines divide washout into an early and late washout with 60 seconds after contrast agent injection. If the lesion present with a completely "black hole" within 2 minutes, it is classified as marked washout, otherwise it is mild washout. The current judgment of the degree of washout is based on the subjective decision made by the observer subjectively, which cannot distinguish the subtle differences in the image and has a subjective dependence. The consistency among the observers is uneven, which affects the diagnostic efficiency of CEUS LI-RADS. Based on this, the purpose of this study was to quantify the key parameters of CEUS LI-RADS: Washout Onset and Washout Degree, and propose standardized and objective diagnostic criteria, to reduce the differences between observers and further improve its diagnostic sensitivity for high-risk groups of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk groups of HCC: patients with liver cirrhosis or chronic viral hepatitis B, or patients who have been diagnosed with HCC or have a history of HCC in the past, as well as adult liver transplant patients and follow-up patients after liver transplantation;
2. CEUS and contrast-enhanced CT/MRI examinations were performed within 2 months before surgery;
3. There are clear surgical pathological or puncture pathological results;
4. Clinical, imaging, and pathological data are complete

Exclusion Criteria:

1. Patients who are not suitable for LI-RADS: patients aged 18 years old or liver cirrhosis caused by congenital liver fibrosis or liver cirrhosis due to hepatovascular disease or diffuse regenerative nodules in the liver;
2. Those who underwent drug therapy (chemotherapy, immunotherapy, and targeted therapy) or local treatment of target lesions (TACE, radiotherapy, radiofrequency ablation, microwave ablation, etc.);
3. The quality of the patient's preoperative image or surgical pathological image is poor or incomplete;
4. Those with annular hyperenhancement or marginal nodular hyperenhancement of arterial lesions in contrast-enhanced ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk groups of HCC with pathology results
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
pathology results | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No